CLINICAL TRIAL: NCT04141943
Title: Improvement of Patient Experience and Healthcare Providers' Productivity Using Virtual Reality in the Field of Radiation Therapy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 4-2019-0795
Record Dates: First submitted 2019-10-21; First posted 2019-10-28 (Actual); Last update posted 2020-11-18 (Actual); Status verified 2020-11

CONDITIONS: Breast Cancer
Keywords: Breast cancer; radiotherapy; virtual reality
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VR (Experimental): The patients who are allocated to the VR arm will receive information about radiotherapy via virtual reality
  Interventions: Other: Virtual reality
- Printed document (No Intervention): The patients who are allocated to the Printed document arm will receive information about radiotherapy via printed document.

INTERVENTIONS:
Other: Virtual reality — The patients who are allocated to the VR arm will receive information about radiotherapy via virtual reality.
  Arms: VR

SUMMARY:
The purpose of this study is to investigate the effect of providing information about radiotherapy using virtual reality and to see whether it would improve the productivity of medical staff, improve patient experience and satisfaction, and reduce patient's anxiety prior to radiotherapy.

DETAILED DESCRIPTION:
All patients enrolled in this study will receive the same routine explanation all radiotherapy patients receive currently. However, prior to the routine explanation, additional detailed information regarding radiotherapy (from simulation to treatment) will be given in two different ways.

VR arm: The patients who are allocated to the VR arm will receive information about radiotherapy via virtual reality.

Printed document arm: The patients who are allocated to the Printed document arm will receive information about radiotherapy via printed document.

Patients will answer the questionnaire related to the anxiety scale related to radiotherapy and measure the vital signs such as blood pressure, pulse rate, and the respiratory rate. Also, patients will answer the questions about radiotherapy to assess the understanding of radiotherapy and questionnaire on hospital satisfaction.

ELIGIBILITY:
Inclusion Criteria:

1. Breast cancer patients who received curative surgery and are planned to receive radiotherapy
2. Patients with cognitive abilities to receive virtual reality information
3. Patients who are 20 years old or older

Exclusion Criteria:

1. Patients who have vision or hearing problems to receive information
2. Patients who do not agree to this study
3. Pregnancy, Fetuses / Newborns, Minors, and Deficient Patients
4. 65 years old or older
5. Patients who have been treated for dizziness within the last 6 months
6. Patients who have experienced severe dizziness within the last 6 months when using electronic devices

Ages: 20 Years to 64 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 196 (Estimated)
Dates: Start 2020-03-13 (Actual); Primary Completion 2021-10 (Estimated); Study Completion 2021-10 (Estimated)

PRIMARY OUTCOMES:
Amsterdam Preoperative Anxiety and Information Scale (APAIS) | Prior to receiving the radiotherapy information via VR or printed document
  Changes in APAIS Before and After Providing Virtual Reality or Printed Document Information
  - APAIS: scale from 1 (not worried at all) to 5 (extremely worried, most anxious)
Amsterdam Preoperative Anxiety and Information Scale (APAIS) | 5 minutes after receiving the radiotherapy information via VR or printed document
  Changes in APAIS Before and After Providing Virtual Reality or Printed Document Information
  - APAIS: scale from 1 (not worried at all) to 5 (extremely worried, most anxious)

SECONDARY OUTCOMES:
State-Trait Anxiety Inventory (STAI) | Prior to receiving the radiotherapy information via VR or printed document
  Changes in STAI Before and After Providing Virtual Reality or Printed Document Information
State-Trait Anxiety Inventory (STAI) | 5 minutes after receiving the radiotherapy information via VR or printed document
  Changes in STAI Before and After Providing Virtual Reality or Printed Document Information

CONTACTS AND LOCATIONS:
Locations (1):
- Severance Hospital, Seoul, Korea, South Korea

IPD SHARING:
Plan to Share IPD: No